CLINICAL TRIAL: NCT06490289
Title: Clinical Efficiency of Psidium Guajava-based Herbal Gel in the Management of Recurrent Aphthous Stomatitis: a Randomized Clinical Trial
Brief Title: Clinical Efficiency of Natural Herbal Based Gel.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Afsheen Mansoor, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2023/43-01
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oral Ulcer
Keywords: Ulcer; Herbel gel
MeSH Terms: conditions — Oral Ulcer; Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Control Group) (No Intervention): No intervention was done
- Group B (Experimental): Denpro oral gel (Gennec Health Sciences PVT, LTD, Karachi, Pakistan) was administered.
  Interventions: Other: Denpro oral gel

INTERVENTIONS:
Other: Denpro oral gel — Experimental group was given Denpro oral gel (Gennec Health Sciences PVT, LTD, Karachi, Pakistan)
  Arms: Group B

SUMMARY:
This clinical trial was conducted in School of Dentistry, Islamabad from 15th June 2023 to 16th January 2024. A total 202 participants took part in study and were divided equally into two groups i.e Control group and Experimental group where Control group was not given any treatment for oral ulcer whereas Experimental group was given herbal based Denpro oral gel 2-4 times a day for at least 4 weeks topically on ulcer area. Mouth ulcer size in patients was measured on first day " Visit=0", second day " Visit=1", third day " Visit=2", fourth day " Visit=3", seventh day " Visit=4" and fourteenth day " Visit=5" for reduction and complete recovery. Data was analyzed by One way ANOVA and POST HOC Tukey test.

DETAILED DESCRIPTION:
This clinical trial was conducted in School of Dentistry, Shaheed Zulfiqar Ali Bhutto medical university for the period of six months from 15th June 2023 to 16th January 2024. Ethical approval was taken from the Ethical Review Board committee of the hospital with the Letter # SOD/ERB/2023/43-01. The participants volunteered in the study after the brief explanation about the aims and objectives study. These participants were enrolled in the study after receiving their informed written consents. Total 202 participants took part in the study and did show up during the entire follow up period of the study. 54 males and 148 females participated in this clinical trial after their confirmation of not having allergy to any type of medication. These patients were divided into two groups i.e Control group and Experimental group. Control group was not given anything but Experimental group was given Denpro oral gel (Gennec Health Sciences PVT, LTD, Karachi, Pakistan) for treating the ulcer 2-4 times a day for at least 2 weeks. They were instructed to apply the gel topically on the ulcer area with the help of finger or applicator after the meals or before sleeping. Moreover, they were forbidden to use any other medication for the treatment of the oral mouth ulcer to avoid the bias. Mouth ulcer size in both the control group and Experimental group was measured on the first day " Visit=0" which was taken as the baseline, again measured on second day " Visit=1" , third day " Visit=2" , fourth day " Visit=3" , seventh day " Visit=4" and finally, fourteenth day " Visit=5". These multiple visits were carried out for checking the reduction in its size and complete recovery of the oral mucosa without using anything in Control group and after the application of the gel in the Experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Mouth ulcer size greater than 2mm that appeared within 48 hours.

Exclusion Criteria:

* Mouth ulcer size lesser than 2mm that did not appear within 48 hours.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Reduction in size of Oral Ulcer and recovery of oral mucosa | treatment of the ulcer 2-4 times a day for at least 2 weeks.
  Mouth ulcer size in both the control group and Experimental group was measured on the first day " Visit=0" which was taken as the baseline, again measured on second day " Visit=1" , third day " Visit=2" , fourth day " Visit=3" , seventh day " Visit=4" and finally, fourteenth day " Visit=5"

CONTACTS AND LOCATIONS:
Overall Officials: Afsheen Mansoor, Ph.D, Principal Investigator — Pakistan Institute of Medical Sciences
Locations (1):
- Afsheen Mansoor, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porter SR, Al-Johani K, Fedele S, Moles DR. Randomised controlled trial of the efficacy of HybenX in the symptomatic treatment of recurrent aphthous stomatitis. Oral Dis. 2009 Mar;15(2):155-61. doi: 10.1111/j.1601-0825.2008.01503.x. PMID 19207485